CLINICAL TRIAL: NCT06826092
Title: Metformin as an Adjunctive Therapy for the Treatment of Metastatic Colorectal Cancer Patients Undergoing FOLFIRI Plus Target Therapy
Brief Title: Metformin for the Treatment of mCRC Patients Undergoing FOLFIRI Plus Target Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jaw-Yuan Wang, MD, PhD, Prof., Kaohsiung Medical University Chung-Ho Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KMUHIRB-F(I)-20220106
Record Dates: First submitted 2025-01-27; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-01

CONDITIONS: Progression-Free Survival
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study group (Experimental): Metformin 500mg TID、FOLFIRI (Leucovorin 200 mg/m2、5-FU 2800 mg/m2、Irinotecan 180 mg/m2) plus target therapy
  Interventions: Drug: Metformin Pill
- Control group (Placebo Comparator): FOLFIRI (Leucovorin (LV), 200 mg/m2, 2-hour infusion, 5-FU, 2,800 mg/m2, 46-hour infusion, Irinotecan (IRI), 180 mg/m2, 2-hour infusion) plus target therapy
  Interventions: Drug: FOLFIRI plus target therapy only

INTERVENTIONS:
Drug: Metformin Pill — Metformin 500mg TID、FOLFIRI (Leucovorin 200 mg/m2、5-FU 2800 mg/m2、Irinotecan 180 mg/m2) plus target therapy
  Other Names: Glucophage
  Arms: Study group
Drug: FOLFIRI plus target therapy only — FOLFIRI (Leucovorin (LV), 200 mg/m2, 2-hour infusion, 5-FU, 2,800 mg/m2, 46-hour infusion, Irinotecan (IRI), 180 mg/m2, 2-hour infusion) plus target therapy
  Arms: Control group

SUMMARY:
To investigate progression-free survival (PFS) in patients with metastatic colorectal cancer treated with chemotherapy FOLFIRI monotherapy or chemotherapy FOLFIRI combined with Metformin

DETAILED DESCRIPTION:
Objectives:

1. Main purpose

   • To investigate progression-free survival (PFS) in patients with metastatic colorectal cancer treated with chemotherapy FOLFIRI monotherapy or chemotherapy FOLFIRI combined with Metformin
2. Secondary purpose (1) To investigate the survival (OS) of patients with metastatic colorectal cancer treated with chemotherapy FOLFIRI monotherapy or chemotherapy FOLFIRI combined with Metformin (2) To investigate the disease control rate (DCR) of patients with metastatic colorectal cancer treated with chemotherapy FOLFIRI monotherapy or chemotherapy FOLFIRI combined with Metformin

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 20 and 90 years old
2. Patients diagnosed with metastatic colorectal cancer who is going to receive FOLFIRI chemotherapy
3. Female must not be planning to become pregnant or breastfeeding, and not pregnant at any point during treatment. (Contraception is required to participate in this trial)
4. Those without major physiological diseases (example of major cardiovascular disease is acute myocardial infarction; example of major cerebrovascular disease is acute stroke, malignant hypertension, acute kidney failure, acute liver failure)
5. Those who are not allergic to the relevant drugs required for the test
6. Those who can follow the doctor's order to take the medicine
7. Subjects must be willing to sign the consent form
8. Blood sugar level above 80 mg/dL

Exclusion Criteria:

Subjects who meet any of the following exclusion conditions are not allowed to join the trial

1. Patients other than the above-mentioned main inclusion criteria.
2. Non-native speakers
3. Known allergy to metformin or any of its components.
4. Severe instability in diabetes (ketoacidosis).
5. Blood sugar level lower than 80 mg/dL
6. Heart failure, respiratory insufficiency.
7. inadequate hematopoietic function defined as below:

   * hemoglobin < 9 g/dL;
   * absolute neutrophil count (ANC) < 1,500/mm3;
   * platelet count < 100,000/mm3;
8. inadequate organ functions defined as below:

   * total bilirubin > 2 times upper limit of normal (ULN);
   * hepatic transaminases (ALT and AST) > 2.5 x ULN;
   * creatinine > 1.5 x ULN;

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-10-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease progression-free survival (PFS) | The trial will continue to follow (approximately every 4 weeks) the subject's survival status until death, loss of follow-up, end of trial, or termination of the trial, assessed up to 52 months
  Disease progression-free survival (PFS) was defined as the date from the initiation of trial treatment until the date of the first imaging-confirmed progression or death (whichever occurred first)

CONTACTS AND LOCATIONS:
Locations (1):
- Chung-Ho Memorial Hospital, Kaohsiung Medical University:, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared. Results will be published by the investigators in academic journals.